CLINICAL TRIAL: NCT05164380
Title: Picture Naming in the Context of Image Type and Response Variety in People With and Without Aphasia
Status: Completed | Type: Observational
Sponsor: Simone Hemm-Ode (Other)
Responsible Party: Sponsor-Investigator, Simone Hemm-Ode, Professor, University of Applied Sciences and Arts Northwestern Switzerland
Organization: University of Applied Sciences and Arts Northwestern Switzerland (Other)
Other Study IDs: Aphasia_ImageType_LangVariety
Record Dates: First submitted 2021-11-18; First posted 2021-12-20 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-12

CONDITIONS: Aphasia
Keywords: aphasia; picture naming; image type; response variety; E-inclusion; word class; naming latency
MeSH Terms: conditions — Aphasia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PWA: Persons with Aphasia
  Interventions: Other: Picture naming tasks
- CG: Control Group healthy adults without aphasia
  Interventions: Other: Picture naming tasks

INTERVENTIONS:
Other: Picture naming tasks — PWA and CG had to name 128 pictures presented on a tablet, in addition to 8 trial images.

SUMMARY:
The observational study aims to investigate the effect of two factors that influence the ease with which aphasic and healthy participants name visual stimuli. The main factors investigated here are the image type of the visual stimulus (drawing or photographic image) and the response variety (standard language vs dialect). The hypothesis is formulated as follows: The image type of the visual stimulus (drawing or photographic image) and the response variety (standard language or dialect) will have an effect on naming correctness and/or naming latencies in people with aphasia within the picture naming test.

The experiment was as follows: Persons with aphasia and healthy participants were presented with objects and verbs depicted as photographs or illustrations on a tablet. All participants were asked to name the depicted term in two different language varieties as correctly and as fast as possible. Answers were recorded synchronously. No feedback should be given to the participants (=no therapy). The results of picture naming were not analyzed patient-specifically in relation to their condition or therapy. Naming performance was collected as a momentary data set in order to investigate the speed of naming in general.

The ethic committee Northwestern and Central Switzerland approved the study to be observational as no effect of intervention(s) on biomedical or other health related outcomes were evaluated, but only the influence of type of the visual stimulus and the response variety on correctness and naming latencies in the two participant groups.

DETAILED DESCRIPTION:
Qulity assurance:

To verify the presence and reliability of all subject data, the following items were checked during these visits using a checklist: Presence of informed consent, presence of all data requested in the questionnaire, correctness of the data copied from the source files (e.g. test protocols) and traceability of the data flow. At the end of the experiment, the correct storage of the data (informed consent of the study participants, identification list, raw data) were checked. All involved staff who had access to the clinical data were informed and trained about anonymization, ethical aspects and correct data manipulation and storage. Direct access to the source data and all relevant documents and records is guaranteed to the ethics committee upon request and presentation.

Data dictionary:

* Questionnaire on personal and health-related information of the experiment participants: Frequencies, descriptive statistics
* The Pyramids and Palm Trees test (PPTT) (Howard & Patterson 1992): passed/not passed: scores above 90% indicate correct cognitive semantics, scores below indicate impaired; 90% of the images must be correctly matched, i.e., at least 47 of 52 items.
* Colouring of Pictures test (CoPT) (De Renzi et al. 1972): passed/not passed: In order to exclude the presence of an acquired color diagnosis due to the brain injury suffered by participants with aphasia, the ability to assign colors to objects is tested with a coloration test.
* Picture Naming Test: Number of correct responses and naming latencies when picture stimuli are presented in two language varieties (Swiss dialect and Swiss standard language)

Data recording and source data:

Case Report Forms (CRF) were printed out on paper and given to experiment participants and practice partners to collect personal and health-related data. Personal and health-related source data was collected in hard copy in the CRF and hard copies were given to study participants and practice partners. Data from pretesting (PPTT, CoPT) for experiment participants with aphasia were recorded manually on the CRF, as were any comments about abnormalities during the course of the study. Data needed for analysis of naming correctness and naming latency (audio and, if consent is given, video data) were collected electronically. Data on naming correctness were also collected on the CRF. The qualitative question-guided interview at the conclusion of data collection was recorded electronically, with accompanying key words noted on the CRF.

AAT scores (from Aachener aphasia test scale) as well as other routinely collected data from patient records of participants with aphasia on the type of aphasia present was manually transferred to the CRF by the speech therapists of the collaborators. The CRFs in paper form are digitized by study staff by scanning and manually transferred to electronic data (filling in Excel lists).

Data protection and data security: confidentiality and encryption The collection, transmission, storage and analysis of health-related personal data of this experiment was carried out in accordance with Art. 5 of the HFV (Humanforschungsgesetz) and in strict compliance with Swiss legal data protection regulations. The project data was kept strictly confidential and was only accessible to authorized personnel who needed the data to fulfill their tasks within the research project. All staff were informed about data protection and confidentiality and were subject to the legal requirements. In the CRF and other project-specific documents, participants were only referred to by a unique identification code, which could only be reconstructed by the participants themselves, but which did not allow any conclusions to be drawn about the participants. The participant identification list as well as the signed informed consents were stored in a secure location at the collaborators and was only transferred to the FHNW after the end of the study, where they will be kept in a safe.

Participant data was collected using an application that was programmed for the experiment under the unique participant identification number only. Other relevant personal and health data was collected in paper form in the CRF. Audio recordings were made of study participants during the naming test and, with the consent of the study participants, they were also filmed; the image and audio sequence were stored in each case. The video recording data was only used for further research, education and training purposes with the prior consent of the experiment participants. All subject-related data was encrypted and stored on the tablet's SD card. The SD card was personally transported to the FHNW by the person conducting the study together with the CRF, where it was handed over to the study director. The information was then decrypted and analyzed on an FHNW computer. The decrypted data was stored securely on three external storage media. One was kept as a backup in the FHNW safe, and two others were used for data analysis at the Academy of Art and Design FHNW and at the School of Education FHNW. These external hard drives were kept securely in safes at the respective institutes when not in use. No original data was stored directly on the FHNW computers. Only the results of the data analysis were stored on other personal computers or secured internal servers. The encryption was managed by the project management. Only a few authorized persons know the key. A list is kept of these persons.

Storage of data:

Data obtained from the research project (raw data sets, analysis results, and anonymized documents) will be archived for at least ten years, protected from access, to ensure scientific sustainability. One hard drive is kept in the FHNW safe, one in appropriately secure locations at the IVK (HGK) and ISP (PH) institutes of the FHNW. Only authorized persons have access. Participant identification lists are destroyed. Should the data be destroyed after a minimum of ten years, all electronic data is deleted and the storage area is securely overwritten. Paper sheets such as the CRF are rendered unusable with the file shredder.

Sample size assessment:

Determining the sample size: The power analysis is based on a simulation. A baseline accuracy (e.g., the percentage correct on stimulus type 1, variety 1) for each of the n virtual participants was first defined.A certain effect size for each of the two factors, stimulus and variety was defined. Both factors are assumed to have an effect as large as an odds ratio of 1.3. This size of odds ratio was used to define the odds for each participant and thus the precision in the other cells of the design. Both effects are analyzed for each simulated data set and then analyzed using a generalized linear mixed-effects model (GLMM) with a binomial distribution of outcomes and a random intercept per participant. Power is calculated as the proportion of simulations for which this statistical model detects an effect of both stimulus type and response variety.

Plan for missing data:

Only those data sets in which participants have completed at least two cells of the design (stimulus type x response variety) are included in the analysis. To counteract dropout of experiment participants - caused by withdrawal of experiment participants, by technical problems in data collection, or by insufficiently collected data - more participants are preemptively recruited than statistically necessary (40 instead of 36 subjects per group) to ensure that there will be enough data to represent an effect, should there be one.

Statistical analysis:

The proportion of correct responses in each cell of the design (stimulus type x response variety) is analyzed using a generalized linear mixed regression model with a binomial distribution of outcomes, including a random intercept estimated for each participant.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria PWA

* Diagnosed with minimal, light or moderate aphasia provoked by a left hemisphere cardiovascular accident
* post-acute or chronic phase with a minimum of six weeks post onset
* Swiss German as first language
* sufficient language comprehension to follow the instructions during the experiment
* attention span of minimum 45 minutes
* no indication for dementia and if any only mild dysarthria and apraxia of speech according to the treating speech therapist
* intact color vision
* normal or corrected to normal vision and hearing

Inclusion Criteria CG

* Swiss German as first language
* No neurological diseases in their health history
* Intact color vision
* Normal or corrected to normal vision and hearing

Exclusion Criteria:

Exclusion Criteria PWA

* Not fulfilling the above inclusion criteria
* Severe aphasia
* Aphasia with an associated disorder in the area of access to semantic object information, as indicated by performance on The Pyramids and Palm Trees Test (PPTT)

Exclusion Criteria CG

-Not fulfilling the above inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: PWA were recruited in cooperation with local speech therapists, hospitals and rehabilitation clinics. CG were recruited via inquiries sent to retiree associations, the researchers' circle of acquaintances as well as by asking relatives of participants with aphasia.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2019-04-29 (Actual); Primary Completion 2021-01-28 (Actual); Study Completion 2021-01-28 (Actual)

PRIMARY OUTCOMES:
Naming correctness | Data were assessed during picture naming test on the test day (upto 1 month after inclusion).
  The degree of correctness or incorrectness of the responses was coded manually following defined criteria. Response of the naming task was considered correct if the participant provided exclusively the previously defined reaction to the stimuli within 10 seconds. To be defined as extended correct response the reaction had to be classified as a synonym or a diminutive of the requested term. Responses describing a generic concept (e.g. "dog" instead of "poodle"), providing too much specification (e.g. rain coat instead of coat) were accounted as extended correct. The same applied for plural forms given instead of singulars.
Naming latencies | Data were assessed during picture naming test on the test day (upto 1 month after inclusion).
  Naming latencies were only calculated for correct responses. Each naming latency was calculated as an interval by measuring the onset of correct target response following after the onset of visual naming stimulus on the tablet screen. Naming latencies were manually measured through using the speech analysis program Praat (Boersma, 2001), which allows acoustic analysis by presenting waveform and spectrogram of audio data.
  Limit: 999 characters.

CONTACTS AND LOCATIONS:
Overall Officials: Simone Hemm-Ode, PhD, Study Chair — University of Applied Sciences Northwestern Switzerland; Institute for Medical Engineering and Medical Informatics
Locations (20):
- Switzerland (20):
  - Kantonsspital Aarau, Aarau
  - Logo Treffpunkt, Altdorf
  - Praxis LogoTreffpunkt, Altdorf
  - Kantonsspital Baden, Baden
  - Felix Platter Spital, Basel
  - REHAB Basel, Basel
  - Kantonsspital Baselland, Liestal
  - Fachhochschule Nordwestschweiz, Muttenz
  - Rundum Therapie, Oberwil
  - Kantonsspital Olten, Olten
  - Praxis für Logopädie, Pratteln
  - Reha Rheinfelden, Rheinfelden
  - Spitäler Schaffhausen, Schaffhausen
  - Privat Klinik im Park Schinznach, Schinznach Bad
  - Rundum Therapie, Therwil
  - Spital Zofingen, Zofingen
  - Logopädische Praxis Dietiker, Zurich
  - Praxis Unterstrass, Zurich
  - Stadtspital Waid, Zurich
  - Universitätsspital Zürich, Zurich

IPD SHARING:
Plan to Share IPD: No